CLINICAL TRIAL: NCT05214222
Title: Penpulimab Plus Chemotherapy With or Without Anlotinib as First-line Therapy for Patients With Advanced Esophageal Squamous Cell Carcinoma (Answer): A Randomized Two-arm Clinical Study
Brief Title: Penpulimab Plus Chemotherapy With/Without Anlotinib for Patients With Advanced Esophageal Squamous Cell Carcinoma
Acronym: ANSWER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2021-405
Record Dates: First submitted 2022-01-03; First posted 2022-01-28 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Advanced Esophageal Squamous Cell Carcinoma
Keywords: PD-1 inhibitor/anlotinib
MeSH Terms: interventions — anlotinib; penpulimab; Paclitaxel; Cisplatin; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Penpulimab plus chemotherapy with Anlotinib
  Interventions: Drug: Anlotinib/Penpulimab/Chemotherapy
- group B (Experimental): Penpulimab plus chemotherapy
  Interventions: Drug: Penpulimab/Chemotherapy

INTERVENTIONS:
Drug: Anlotinib/Penpulimab/Chemotherapy — Initial treatment (4-6 cycles): Anlotinib, Penpulimab, Paclitaxel or Albumin Paclitaxel,Cisplatin
  * Anlotinib: once a day, 1 capsule each time (10mg for body weight <60KG, 12mg for body weight ≥60KG), d1-d14, 3 weeks as a treatment cycle.
  * Penpulimab: 200 mg, d1 per cycle, once every 3 weeks.
  * Paclitaxel: According to 135-175mg/m2, intravenous infusion> 2h, d1, 3 weeks as a treatment cycle; Albumin paclitaxel: According to 200-260mg/m2, intravenous infusion for 30 minutes, d1, 3 weeks as a treatment cycle.
  * Cisplatin: 60-75mg/m2, intravenous infusion, divided into d1-d3 medication per cycle; 3 weeks is a treatment cycle.
  Maintenance treatment: Anlotinib, Penpulimab
  * Anlotinib: once a day, 1 capsule each time (the same as the initial treatment dose), take the drug every cycle d1-d14, 3 weeks as a treatment cycle.
  * Penpulimab: 200mg, d1 per cycle, once every 3 weeks
  Other Names: Anlotinib, Penpulimab, Paclitaxel or Albumin Paclitaxel,Cisplatin
  Arms: group A
Drug: Penpulimab/Chemotherapy — Initial treatment (4-6 cycles): Penpulimab, Paclitaxel or Albumin Paclitaxel,Cisplatin
  * Penpulimab: 200 mg, d1 per cycle, once every 3 weeks.
  * Paclitaxel: According to 135-175mg/m2, intravenous infusion> 2h, d1, 3 weeks as a treatment cycle; Albumin paclitaxel: According to 200-260mg/m2, intravenous infusion for 30 minutes, d1, 3 weeks as a treatment cycle.
  * Cisplatin: 60-75mg/m2, intravenous infusion, divided into d1-d3 medication per cycle; 3 weeks is a treatment cycle.
  Maintenance treatment: Penpulimab
  • Penpulimab: 200mg, d1 per cycle, once every 3 weeks Post-progression genetic testing, continued treatment: Anlotinib,Penpulimab Anlotinib: Once daily, one capsule per time (10mg for weight <60KG, 12mg for weight ≥60KG), administered from day 1 to day 14 of each cycle. Two consecutive weeks of treatment followed by one week off, 3 weeks per treatment cycle.
  Penpulimab: 200mg, administered on day 1 of each cycle, every 3 weeks.
  Other Names: Penpulimab, Paclitaxel or Albumin Paclitaxel,Cisplatin
  Arms: group B

SUMMARY:
Penpulimab plus chemotherapy with or without Anlotinib as first-line therapy for patients with advanced esophageal squamous cell carcinoma (Answer): A randomized two-arm clinical study.

DETAILED DESCRIPTION:
This is a open-label, phase II study of Penpulimab plus chemotherapy with or without Anlotinib as first-line therapy in subjects With resectable advanced esophageal squamous cell carcinoma. The patients will be divided into two groups. In group A, Penpulimab plus chemotherapy with Anlotinib will be given every 3 weeks for 4-6 cycles in initial stage, then in maintenance treatment, Anlotinib and Penpulimab will be used every 3 weeks until disease progression or intolerance; In group B, Penpulimab plus chemotherapy will be given every 3 weeks for 4-6 cycles in initial stage, then penpulimab will be used every 3 weeks until disease progression, Anlotinib and Penpulimab will be used every 3 weeks until disease progression again or intolerance;

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage III-IV esophageal squamous cell carcinoma who are not candidates for curative treatment (excluding adenosquamous carcinoma mixed type);
2. Those who have not received systemic treatment in the past, or (new) adjuvant treatment/radical surgery/radical radiotherapy and chemotherapy have relapsed for more than 6 months; Note: Including patients with advanced or recurring non-target lesions who have progressed again after radiotherapy alone. For local lesions (non-target lesions), the time from the end of palliative treatment to the enrollment time> 2 weeks;
3. According to the RECIST 1.1 version of the curative effect evaluation standard for solid tumors, there is at least one measurable lesion; the measurable lesion should not have received local treatment such as radiotherapy (the lesion located in the previous radiotherapy area, if it is confirmed that it has progressed, and meets RECIST1.1 Standard, target lesions can also be selected);
4. Patients between 18 and 75 years old;
5. ECOGPS score: 0~1 points; the expected survival period is more than 3 months;
6. Tumor specimens can be provided to determine gene detection and PD-L1 expression, at least 15 white sheets (assessed by the company); provide two oral swabs; within 7 days before the medication, the first, third, and sixth at the end of the cycle, one tube of 6ml EDTA anticoagulant blood will be provided.
7. It has sufficient organ and bone marrow function, that is, it meets the following standards:

(1) The standard of routine blood examination must meet: Hemoglobin content (HB) ≥90g/L (no blood transfusion within 28 days); Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥100×10^9/L. (2) The biochemical inspection shall meet the following standards: Serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); ALT and AST≤2.5´ULN; if there is liver metastasis, ALT and AST≤5´ULN; Cr≤1.5´ULN or creatinine clearance (CCr)≥60ml/min; (Cockcroft-Gault formula) (3) The coagulation function is adequate, which is defined as the international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; 8) Women of childbearing age must take appropriate contraceptive measures from screening to 3 months after stopping the treatment, and they must be non-lactating patients. Before starting the administration, the pregnancy test is negative, or meeting one of the following criteria proves that there is no risk of pregnancy:

1. Post-menopausal is defined as amenorrhea at least 12 months after the age is greater than 50 years and all exogenous hormone replacement therapy is stopped;
2. For women younger than 50 years old, if the amenorrhea is 12 months or more after stopping all exogenous hormone treatments, and the levels of luteinizing hormone (LH) and follicle stimulating hormone (FSH) are within the laboratory postmenopausal reference value range, also Can be considered post-menopausal;
3. Have received irreversible sterilization, including hysterectomy, bilateral ovariectomy or bilateral fallopian tube resection, except for bilateral tubal ligation.

For men, they must agree to use appropriate methods of contraception or have been surgically sterilized during the trial period and 8 weeks after the last trial drug administration; 9) The patient voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. It is known that esophageal squamous cell carcinoma tends to be completely obstructed under endoscopy and requires interventional treatment to relieve the obstruction;
2. Patients with ulcerative esophageal squamous cell carcinoma;
3. Patients who have a higher risk of bleeding or perforation due to the tumor's obvious invasion of the adjacent organs (aorta or trachea) of the esophageal lesion, or patients who have formed a fistula;
4. Patients with esophageal squamous cell carcinoma whose esophageal lesions have not been reduced after radiotherapy without surgical resection of the primary lesion;
5. Allergy to paclitaxel and cisplatin preparations or excipient ingredients;
6. Patients who have used paclitaxel or cisplatin in adjuvant chemotherapy and have relapsed or metastasized within six months; Note: Those who have relapsed or metastasized for more than six months can be included in the study;
7. Previously received anti-tumor immunotherapy (including immune checkpoint inhibitors, immune cell therapy, etc.) or anti-angiogenesis targeted therapy drugs (including antibodies and small molecule tyrosine kinase inhibitors);
8. There are many factors that affect oral medications (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), but patients who have difficulty swallowing and can drink, can take Anlotinib after dissolving the granules;
9. The burden of liver metastases accounts for more than 50% of the entire liver volume;
10. Patients with any severe and/uncontrolled diseases, including:

    1. Patients with unsatisfactory blood pressure control using antihypertensive drugs (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg); patients with grade II or higher myocardial ischemia or myocardial infarction, arrhythmia (including QT interval ≥480ms); according to NYHA standards , Grade III-IV cardiac insufficiency, or cardiac color Doppler ultrasound examination reveals that the left ventricular ejection fraction (LVEF) is less than 50%;
    2. Active or uncontrolled serious infection;
    3. Liver diseases such as cirrhosis, decompensated liver disease, chronic active hepatitis;
    4. Poor control of diabetes (fasting blood glucose (FBG)> 10mmol/L);
    5. Urine routines suggest that urine protein is ≥++, and the 24-hour urine protein content is confirmed to be greater than 1.0g;
11. Long-term unhealed wounds or fractures;
12. Patients with esophageal squamous cell carcinoma with active bleeding within 2 months of the primary lesion; pulmonary hemorrhage with NCICTCAE grade> grade 1 occurred within 4 weeks before enrollment; other sites with NCICTCAE grade> grade 2 occurred within 4 weeks before enrollment Bleeding; patients with bleeding tendency (such as active peptic ulcer) or who are receiving thrombolytic or anticoagulant therapy such as warfarin, heparin or their analogues;
13. Major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks before the first dose of the study or expected major surgery during the study treatment period.
14. A history of gastrointestinal perforation and/or fistula in the 6 months before the enrollment treatment; or arteriovenous thrombotic events, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and lungs Embolizer
15. There are known symptomatic central nervous system metastases and/or cancerous meningitis;
16. Ascites with clinical significance, including any ascites that can be found on physical examination, ascites that has been treated in the past or still needs to be treated at present, only those with a small amount of ascites but asymptomatic on imaging can be selected;
17. Patients with moderate pleural effusion on both sides, or large pleural effusion on one side, or patients who have caused respiratory dysfunction and require drainage;
18. Known to have active tuberculosis;
19. Suffer from interstitial lung disease that requires steroid therapy;
20. Uncontrolled metabolic disorders or other non-malignant tumor organs or systemic diseases or cancer secondary reactions, which may lead to higher medical risks and/or uncertainty in survival evaluation;
21. Patients with significant malnutrition, BMI<13.6kg/m2;
22. People who have a history of psychotropic drug abuse and cannot be quit or have mental disorders;
23. Have a history of immunodeficiency, including those who have tested positive for HIV or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
24. History of other primary malignant tumors, except for the following: 1) Malignant tumors that have been completely remitted for at least 2 years before enrollment and no other treatment is required during the study period; 2) Non-melanoma skin that has been adequately treated and has no evidence of disease recurrence Carcinoma or malignant freckle-like nevus; 3) Carcinoma in situ that has been adequately treated and has no evidence of disease recurrence;
25. Female patients who are pregnant or breastfeeding;
26. According to the judgment of the investigator, those with concomitant diseases that seriously endanger the safety of the patient or affect the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2028-09-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to approximately 2 year
  ORR was defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to approximately 2 year
  DCR was defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) or a Stable Response per RECIST 1.1
Progression Free Survival (PFS) include PFS1,PFS2 | up to approximately 2 year
  PFS was defined as the time from first day of study treatment to the first documented PD or death due to any cause during the specific treatment period, whichever occurred first
Overall Survival (OS) | up to approximately 3 year
  OS was defined as the time from first day of study treatment to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up
Safety: AE | up to approximately 2 year
  Safety was defined as the Number of Participants With an Adverse Event
Change From Baseline in Health-related Quality of life (HRQoL) Score Using European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) | up to approximately 2 year
  The EORTC QLQ-C30 is a questionnaire to assess the overall HRQoL. Participant responses to the question " How would you rate your overall quality of life (QoL) during the past week?" are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall QoL. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in HRQoL EORTC QLQ-C30 score in participants will be presented.
Change From Baseline in HRQoL Score Using EORTC Quality of Life Questionnaire-Oesophageal Module (QLQ-OES18) | up to approximately 2 year
  The EORTC QLQ-OES18 is a disease-specific questionnaire to assess measurements specific to esophageal cancer. It contains 18 items and is based on four subscales-dysphagia, eating, reflux and pain. All items are scored using a four-point scale that offers these response choices: 1=not at all, 2=a little, 3=quite a bit, 4=very much. A higher score indicates worse level of symptoms. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in HRQoL QLQ-OES18 score in participants will be presented.
The 1-year OS rate | 1 year
  OS was defined as the time from first day of study treatment to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up
The 2-year OS rate | 2 years
  OS was defined as the time from first day of study treatment to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up
The 3-year OS rate | 3 years
  OS was defined as the time from first day of study treatment to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: wei wang, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China